CLINICAL TRIAL: NCT03732950
Title: A Phase II Study of Pembrolizumab Monotherapy in Recurrent Ovarian Cancer of the Immunoreactive Subtype Determined by NanoString Gene Expression Profiling
Brief Title: Pembrolizumab in Treating Participants With Recurrent Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000643; NCI-2018-01550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-000643 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Participants receive pembrolizumab intravenously IV on day 1. Courses repeat every 3 weeks for up to 35 courses (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating participants with ovarian cancer that has come back after previous treatment. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate clinical anti-tumor activity of pembrolizumab monotherapy based on objective response rate (ORR) as assessed by the investigator per immune related Response Evaluation Criteria in Solid Tumors (irRECIST) in patients with recurrent ovarian cancer (ROC) whose tumors show an immunoreactive gene expression signature.

SECONDARY OBJECTIVES:

I. To evaluate clinical anti-tumor activity of pembrolizumab monotherapy based on progression-free survival (PFS) as assessed by the investigator per irRECIST in patients with ROC whose tumors show an immunoreactive gene expression signature.

II. To evaluate clinical anti-tumor activity of pembrolizumab monotherapy based on PFS rate at 6, 12 and 18 months as assessed by the investigator per irRECIST in patients with ROC whose tumors show an immunoreactive gene expression signature.

III. To evaluate and characterize the tolerability and safety profile of the study population after being treated with pembrolizumab as monotherapy.

EXPLORATORY OBJECTIVES:

I. To assess correlations of the immunoreactive gene signature with the validated a PD-L1 immunohistochemistry (IHC) assay using Merck's proprietary 22C3 antibody and the clinical activity observed in the study population.

OUTLINE:

Participants receive pembrolizumab intravenously (IV) on day 1. Courses repeat every 3 weeks for up to 35 courses (2 years) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 and then every 9 and 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have received 1-5 prior lines for treating ROC (i.e. 2-6 total prior lines counting the front line) and must have a platinum-free interval (PFI) or a treatment-free interval (TFI) >= 3 months based on the last regimen received
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

  * Note: Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Have histologically diagnosed recurrent epithelial ovarian, fallopian or primary peritoneal ovarian cancer
* Have provided a tumor tissue sample either collected from a newly obtained tumor tissue biopsy or an archival tissue specimen. Subjects for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived biopsy specimen. Formalin-fixed paraffin embedded (FFPE) block specimens are preferred to 20 unstained slides. Additional samples may be requested if tumor tissue provided is not adequate for quality and/or quantity as assessed by the central laboratory
* Performed within 10 days of treatment initiation: absolute neutrophil count (ANC) >= 1,500/mcL
* Performed within 10 days of treatment initiation: platelets >= 100,000/mcL
* Performed within 10 days of treatment initiation: hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Performed within 10 days of treatment initiation: serum creatinine OR measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) =< 1.5 x upper limit of normal (ULN) OR >= 45 mL/min for subject with creatinine levels > 1.5 x institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Performed within 10 days of treatment initiation: serum total bilirubin =<1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Performed within 10 days of treatment initiation: aspartate aminotransferase (AST) (serum glutamate pyruvate transaminase [SGOT]) and aspartate aminotransferase (ALT) (serum glutamic-oxaloacetic transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Have received front line platinum-based chemotherapy (preoperative chemotherapy is allowed)
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2025-03-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed per immune related Response Evaluation Criteria in Solid Tumors (irRECIST) | Up to 2 years
  ORR will be calculated with corresponding 95% unadjusted exact binomial confidence interval (CI).

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed per irRECIST | At 6, 12, and 18 months
  The Kaplan?Meier method will be used to summarize PFS and PFS at 6 months.
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Konecny, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota